CLINICAL TRIAL: NCT01760668
Title: Aortopathy in Persons With Bicuspid Aortic Valve, Turner and Marfan Syndrome
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 1-10-72-561-12
Record Dates: First submitted 2013-01-02; First posted 2013-01-04 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2015-06

CONDITIONS: Turner Syndrome; Bicuspid Aortic Valve; Marfan Syndrome
Keywords: Sex chromosome; Turner Syndrome; Marfan syndrome; Bicuspid aortic valve; Aortic Aneurysm; Epigenetics; Transcriptome; non-coding RNA; Electron microscopy; Proteomics
MeSH Terms: conditions — Turner Syndrome; Bicuspid Aortic Valve Disease; Marfan Syndrome; Aortic Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Aortic tissue
  Blood Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Turner syndrome (TS): TS verified by genotyping Age > 18 years awaiting operation due to aortic dilation
- Marfan syndrome (MS): Females with MS verified clinically or by genotyping Age > 18 years awaiting operation due to aortic dilation
- Bicuspid aortic valve: females with bicuspid aortic valve Age > 18 years awaiting operation due to aortic dilation
- Controls: Men/females who died from conditions other than aortic dilation or dissection. Age 20-60 years.

SUMMARY:
The study aim is:

1. To examine aortic tissue by light microscopy
2. To examine aortic tissue by electron microscopy
3. To study changes in the epigenome and transcriptome of the X chromosome specific to aortic tissue.
4. To examine aortic tissue using biochemistry including proteomics.
5. To establish the karyotype of fibroblasts with standard chromosome examination on 10 meta-phases as well as by fluorescent in situ hybridization (FISH) with probes covering the X and Y chromosome. Using the latter 200 meta-phases will be examined.

30 controls who did not die from aortic dissection or dilation will be recruited from The Department of Forensic Medicine at Aarhus University Hospital.

The investigators will subject samples of aortic tissue from women undergoing prophylactic aortic surgery due to either Marfan syndrome or bicuspid aortic valve to the same panel of examinations (except karyotyping). Lastly the investigators will compare the results from the three groups (Turner syndrome, Marfan syndrome and Bicuspid aortic valve).

DETAILED DESCRIPTION:
Turner syndrome is a congenital complete or partial lack of one of the female sex chromosomes affecting 1 of 2000 live born girls. The syndrome is characterized by an increased prevalence of ischemic heart disease, aortic dilation and dissection, hypertension, stroke and autoimmune diseases in general.

ELIGIBILITY:
Turner syndrome (TS).

A. Inclusion

* TS verified by genotyping
* Age > 18 years
* Awaiting operation due to aortic dilation

B. Exclusion - Previous aortic dissection or operation of the aorta (per-cutaneous or open surgery)

Marfan syndrome (MS)

A. Inclusion

* Females with MS verified clinically or by genotyping
* Age > 18 years
* Awaiting operation due to aortic dilation

B. Exclusion

- Previous aortic dissection or operation of the aorta (per-cutaneous or open surgery)

Bicuspid aortic valve

A. Inclusion

* Females with Bicuspid aortic valve
* Age > 18 years
* Awaiting operation due to aortic dilation

B. Exclusion - Previous aortic dissection or operation of the aorta (per-cutaneous or open surgery)

Controls

A. Inclusion

* Men/females who died from conditions other than aortic dilation or dissection.
* Age 20-60 years.

B. Exclusion

- Previous aortic dissection or operation of the aorta (per-cutaneous or open surgery)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with Turner syndrome will be recruited from out-patient clinics. Individuals with Turner syndrome, Marfan syndrome and bicuspid aortic valve will be recruited from departments of cardiology or thoracic surgery in Odense, Copenhagen or Aarhus (Denmark).
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2013-02; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Histone modifications | Cross sectional
  Permissive and repressive histone modifications on the X-chromosome
mRNA and non-coding RNAs | Cross sectional
  Identification of the entire transcriptome including both mRNA and non-coding RNAs (lincRNA as well as miRNA)from the X-chromosome
DNA-methylations of CpG-islands | Cross sectional
  mapping DNA-methylations of CpG-islands
Electron microscopic evaluation | Cross sectional
Karyotyping by FISH and conventional karyotyping | Cross sectional
Proteomics | Cross sectional

CONTACTS AND LOCATIONS:
Overall Officials: Christian Trolle, Principal Investigator — Aarhus University Hospital; Claus H Gravholt, MD, Ph.d., Study Director — Aarhus University Hospital
Locations (1):
- Department of Endocrinology and Internal medicine, Aarhus C, Denmark